CLINICAL TRIAL: NCT01734694
Title: Safety and Efficacy of Strategy to Prevent Drug-Induced Nephrotoxicity in High-Risk Patients
Acronym: STOP-NT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Independent biostatistician recommended early termination of the trial due to low probability of success.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Jose Vazquez, M.D., Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7089
Record Dates: First submitted 2012-11-14; First posted 2012-11-28 (Estimated); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Health Care Associated Pneumonia; Osteomyelitis/Septic Arthritis; Endocarditis; Bacteremia; Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: conditions — Osteomyelitis; Arthritis, Infectious; Endocarditis; Bacteremia | interventions — Vancomycin; Ceftaroline; Daptomycin; Linezolid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin
- Comparator (Active Comparator)
  Interventions: Drug: Ceftaroline; Drug: Daptomycin; Drug: Linezolid

INTERVENTIONS:
Drug: Vancomycin — Dose optimized vancomycin. Target trough: 15 - 20 mg/L for Health Care Associated Pneumonia, Osteomyelitis, Septic Arthritis, Endocarditis and Bacteremia;
  Target trough: 10 - 20 mg/L for Acute Bacterial Skin and Skin Structure Infections;
  Arms: Vancomycin
Drug: Ceftaroline — Dose based on package insert labeling
  CrCL > 50 mL/min: 600 mg IV q12h
  CrCL 31-50 mL/min: 400 mg q12h
  CrCL 15-30 mL/min: 300 mg q12h
  CrCL < 15mL/min: 200 mg q12h;
  Other Names: Teflaro
  Arms: Comparator
Drug: Daptomycin — Dose based on renal function and literature dosing recommendations
  CrCL ≥ 30 mL/min: 6 - 10 mg/kg IV q24h
  CrCL < 30 mL/min: 6 - 10 mg/kg IV q48h
  Other Names: Cubicin
  Arms: Comparator
Drug: Linezolid — 600 mg IV/PO q12h
  Other Names: Zyvox
  Arms: Comparator

SUMMARY:
For more than fifty years, vancomycin has been cited as a nephrotoxic agent. Reports of vancomycin induced kidney injury (a.k.a vancomycin induced nephrotoxicity or VIN), have waxed and waned throughout the years for various reasons. Recently, VIN has reemerged as a clinical concern. This may be due to various reasons, including new dosing recommendations as well as an increased prevalence of risk factors associated with vancomycin induced nephrotoxicity. This study aims to evaluate a strategy which attempts to reduce kidney damage from vancomycin use.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Receiving intravenous vancomycin for the treatment of healthcare associated pneumonia, osteomyelitis/septic arthritis, endocarditis/bacteremia, or acute bacterial skin and skin structure infections
* Expected to receive vancomycin for at least 72 hours and are within the first 72 hours of therapy
* Have at least two or more of the following risk factors for drug-induced nephrotoxicity: a) receipt high-dose vancomycin therapy (greater than or equal to four grams per day) b) receipt of vasopressors c) receipt of nephrotoxic drugs (i.e. aminoglycosides, furosemide, acyclovir, amphotericin b, colistin, and intravenous contrast dye) d) pre-existing renal dysfunction (i.e. SCr greater than or equal to 1.5 mg/dL).

Exclusion Criteria:

* Pregnancy
* End-stage renal disease
* Receipt of more than 4 grams of vancomycin prior to enrollment on current admission
* Absolute neutrophil count < 1000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Vazquez, M.D., Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator: Ceftaroline: Dose based on package insert labeling
  CrCL > 50 mL/min: 600 mg IV q12h
  CrCL 31-50 mL/min: 400 mg q12h
  CrCL 15-30 mL/min: 300 mg q12h
  CrCL < 15mL/min: 200 mg q12h;
  Daptomycin: Dose based on renal function and literature dosing recommendations
  CrCL ≥ 30 mL/min: 6 - 10 mg/kg IV q24h
  CrCL < 30 mL/min: 6 - 10 mg/kg IV q48h
  Linezolid: 600 mg IV/PO q12h
Period: Overall Study
Arm/Group | Vancomycin | Comparator
Started | 51 | 49
Completed | 51 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin | Comparator | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [51 to 68] | 60 [51 to 68] | 60 [53 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 34 | 29 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 16 | 33
  African American | 32 | 32 | 64
  Hispanic | 1 | 0 | 1
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Individuals With Nephrotoxicity
Description: Increase in SCr of 0.5 mg/dL or 50% above baseline for at least two consecutive days while on the study drug and through discharge from hospital.
  This measure will be reported as proportion of patients with nephrotoxicity within each group in relation to the number of patients in each group.
Time Frame: Day 1 and daily serum creatinine assessment up to date of discharge from hospital, and a median of 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Comparator
Number analyzed (Participants) | 51 | 49
Participants | 5 | 3

2. Secondary Outcome: Proportion of Individuals With Acute Kidney Injury Network Modified Definition of Nephrotoxicity
Description: An abrupt (within 48 hour) reduction in kidney function with one or more of the following 1) Increase in SCr ≥ 0.3 mg/dL 2) Increase SCr ≥ 50% or 3) Decreased urine output (< 0.5 ml/kg/hr x 6 hrs) while on the study drug.
  This measure will be reported as proportion of patients with acute kidney injury within each group in relation to the number of patients in each group.
Time Frame: Day 1 and daily serum creatinine assessment up to date of discharge, and a median of 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Comparator
Number analyzed (Participants) | 51 | 49
Participants | 16 | 16

3. Secondary Outcome: Proportion of Individuals With Clinical Success
Description: Clinical success is a composite endpoint of those patients with clinical cure or improvement in clinical signs and symptoms of infection (i.e. SIRS criteria, and microbiology) while on the study drug.
  This measure will be reported as the proportion of patients with clinical success in each group compared to the the total number of patients in the group.
Time Frame: Daily assessment of signs and symptoms of infection, and a median of 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Comparator
Number analyzed (Participants) | 51 | 49
Participants
  Clinical Success | 42 | 44
  Indeterminate | 4 | 3
  Clinical Failure | 5 | 2

ADVERSE EVENTS:
Arm/Group | Vancomycin | Comparator
Serious Adverse Events (participants affected / at risk) | 16/51 | 16/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vancomycin (N=51) | Comparator (N=49)
Nephrotoxicity (Renal and urinary disorders) | 5 | 3 — Increase in SCr of at least 0.5 mg/dL or 50% (whichever is greater) on at least 2 consecutive measurements while on the study drug.
Acute Kidney Injury (Renal and urinary disorders) | 16 | 16 — An abrupt change in renal function signified by an increase in SCr of at least 0.3 mg/dL, a reduction in creatinine clearance (CrCl) of at least 50%, or a change in urine output to <0.5 mL/kg/h for at least 6 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No